CLINICAL TRIAL: NCT04818606
Title: Mindfulness-Oriented Recovery Enhancement in the Management of Lumbosacral Radiculopathy Symptoms: A Randomized Controlled Trial
Brief Title: MORE in the Management of Lumbosacral Radiculopathy Symptoms: A Randomized Controlled Trial
Acronym: MORE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Natural Medicine (Other)
Responsible Party: Principal Investigator, Katie Pickworth, Adjunct Faculty, National University of Natural Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KP112720
Record Dates: First submitted 2021-03-09; First posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Lumbar Radiculopathy
Keywords: lumbar radiculopathy; Mindfulness Oriented Recovery Enhancement(MORE); mindfulness; integrative and complementary health
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Intervention Model Description: Control Group = treatment as usual (TAU) Intervention Group = 8-week virtual mindfulness session
Who Masked: Investigator, Outcomes Assessor
Masking Description: RAs recruited onto the study team to conduct study visits will not have access to information regarding participant group assignment. Study leads providing the intervention will have the opportunity to run baseline participant visits but will not be allowed to run follow-up study visits for participants in any cohort to which they have delivered an intervention. The Principal Investigator and statistician will be completely blinded to group assignments
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (MORE) Group (Experimental): Participants randomized to the intervention group will undergo an eight-week mindfulness training program as instructed by MORE for the Treatment of Chronic Pain manual. This eight-week intervention will consist of weekly synchronous video conferencing sessions during which participants will be asked to follow along with a guided meditation read by the study lead and to engage in reflection and discussion exercises with other study participants. Participants will also be asked to complete weekly activities and daily mindfulness practices outside of weekly synchronous meetings. Pre-recorded guided meditations created by study personnel using scripts from the MORE manual will be provided to participants to facilitate their daily practice.
  Interventions: Other: Mindfulness Oriented Recovery Enhancement
- Control Group (No Intervention): This group will undergo treatment as usual (TAU) over the course of the eight-week time period of parallel group comparison. This may or may not involve regularly scheduled, standard visits with other medical personnel, including primary care, specialized medical services, or complementary and integrative health practitioners (e.g., acupuncture). Participants will be asked to refrain from altering therapeutic approaches to pain management during this time unless medically necessary and will be asked to report any changes made to their treatment plan on a daily basis.

INTERVENTIONS:
Other: Mindfulness Oriented Recovery Enhancement — Participants randomized to the intervention group will undergo an eight-week mindfulness training program as instructed by MORE for the Treatment of Chronic Pain manual. This eight-week intervention will consist of weekly synchronous video conferencing sessions during which participants will be asked to follow along with a guided meditation read by the study lead and to engage in reflection and discussion exercises with other study participants. Participants will also be asked to complete weekly activities and daily mindfulness practices outside of weekly synchronous meetings.
  Other Names: MORE
  Arms: Intervention (MORE) Group

SUMMARY:
INTRODUCTION: Chronic low back pain (CLBP) is a ubiquitous musculoskeletal (MSK) complaint that often presents as a chronic and difficult to treat condition. Lumbosacral radiculopathy/radiculitis (LR) or "sciatica" is a common secondary condition that can last well beyond the expected time frame after treatment with physical therapy, oral anti-inflammatory medications, local steroidal injections, and surgery. Challenges in the treatment of LR indicate that persistent pain may have evolved from mechanical to neuropathic. Previous research has shown that, in addition to the aforementioned treatments, mindfulness-based stress reduction (MBSR) is effective in limiting self-reported pain in patients with CLBP and neurogenic conditions such as fibromyalgia. This study proposes a randomized clinical trial to evaluate the effects of a newer mindfulness program, Mindfulness Oriented Recovery Enhancement (MORE), on self-reported pain, physical function, quality of life (QoL), depression symptoms, trait mindfulness, reinterpretation of pain, and surface electromyography (sEMG) findings in patients with LR.

METHODS: Participants will be recruited from the Portland, OR metro area. Upon screening and recruitment, participants will receive a battery of questionnaires collecting demographic, self-reported pain, physical function, QoL, depression symptoms, mindfulness, and reinterpretation of pain data. Participants will also undergo sEMG to identify neurological abnormalities that can be characterized diagnostically. Upon enrollment, participants will be randomized to either the mindfulness-based intervention group (MBI), MORE; or the control group, treatment as usual (TAU), for 8 weeks. Self-reported pain measures and sEMG studies will be conducted again at eight weeks post randomization.

HYPOTHESES: Primarily, investigators hypothesize that MORE will be effective in improving self-reported pain, physical function, QoL, depression symptoms, mindfulness, and reinterpretation of pain scores after eight weeks of mindfulness training. Secondarily, investigators hypothesize that those individuals with abnormal sEMG findings at baseline will have improved sEMG findings at their eight-week follow-up visit.

ANALYSIS PLAN: Changes in self-reported pain, physical function, QoL, depression symptoms, trait mindfulness, and reinterpretation of pain will be analyzed using descriptive statistics as well as ANCOVA. Regression will also be used to evaluate the dose-response relationship between all outcome measures and time spent in mindfulness practice for the intervention group. Finally, ANCOVA will be used to evaluate the relationship between pain and physical function and sEMG findings.

ELIGIBILITY:
Inclusion Criteria:

1: Presence of previous diagnosis of LR

1a: Presence of lumbosacral radiculopathy/radiculitis symptoms that extend below the knee secondary to low back pain for greater than 6 weeks with a painDETECT score greater than 18 OR.

1b: Diagnosis of lumbosacral radiculopathy/radiculitis secondary to low back pain that extends below the knee, with symptoms present for greater than 6 weeks.

1b.1: ICD-10 codes used for diagnostic inclusion: M54.16, M54.17, M51.16, M51.17, M47.26, M47.27, M54.40, M54.41, M54.42, M99.53, M99.54, S34.21, S34.22, G54.4, and G55

2: At least 18 years of age and not older than 64 at the time of study enrollment.

3: Ability to read and understand English.

4: Willingness to be randomized to either an experimental or a control group.

5: Willingness to refrain from unnecessary or self-directed pain management/treatment plan changes during study enrollment and to report necessary changes made.

6: Daily access to the internet via cell phone, tablet, or computer.

Exclusion Criteria:

1. Epidural steroid injection in the prior 3 months.
2. Inability to complete 20 unassisted gait cycles.
3. Have received a surgical intervention for low back pain or lumbosacral radiculopathy/radiculitis within the previous 6 months.
4. Current active mindfulness meditation practice: 1 time/week or more and/or formal training in mindfulness/meditation practice.
5. Concurrent diagnosis of cancer.
6. Allergy or intolerance to adhesive.
7. Current unmanaged or uncontrolled mental illness known to cause psychosis: schizophrenia and schizotypal disorders, bipolar I disorder with psychosis, major depressive disorder with psychosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Change in Modified Oswestry Low Back Pain Disability Questionnaire Score | Change from Baseline to 8-Week Follow-Up
  The ODI is designed to assess the intensity of pain and the degree to which pain interferes with activities of daily living such as personal care, lifting, walking, sitting, etc.

SECONDARY OUTCOMES:
Change in painDETECT Questionnaire Score | Change from Baseline to 8-Week Follow-Up
  The PD-Q is a self-reporting pain questionnaire that is designed to assess the presence of neuropathic pain in patients with chronic low back pain and lumbosacral radiculopathy/radiculitis. The PD-Q is scored on a scale from -1 to 38 where scores 19 or greater indicate likely presence of neuropathic pain, scores from 12 to 18 represent ambiguous pain, and scores below 12 represent a likelihood that neuropathic pain is not present.
Change in Visual Analog Scale Score | Change from Intervention Week 1 to Intervention Week 8
  he VAS is a self-reporting scale where participants are asked to report their pain on a scale of 1 to 10 where 0 represents "no pain" and 10 represents "worst pain".
Change in SF-12 Patient Questionnaire for Quality of Life Score | Change from Baseline to 8-Week Follow-Up
  The SF-12 QoL assesses an individual's overall quality of life using self-reporting questions to determine an individual's ability to accomplish and complete activities of daily living as well as their overall mood and outlook on life
Change in Major Depression Inventory Score | Change from Baseline to 8-Week Follow-Up
  The MDI is a self-report questionnaire that includes questions about depression symptoms consistent with the DSM V guidelines for major depressive disorder.
Change in Five Facet Mindfulness Questionnaire Score | Change from Baseline to 8-Week Follow-Up
  The FFMQ is a self-reported questionnaire that assesses an individual's trait mindfulness using five "facets" or categories of mindfulness: Observing, Describing, Acting with Awareness, Nonjudging of inner experience, and Nonreactivity to inner experience. Participants respond to 39 questions such as "I can easily put my beliefs, opinions, and expectations into words" on a scale of never or very rarely true (1) to very often or always true (5).
Change in Mindful Reinterpretation of Painful Sensations Scale Score | Change from Baseline to 8-Week Follow-Up
  he MRPS is a 9 item survey that asks participants to respond to questions regarding their perspective of their pain such as "I try to watch my pain from a distance, as if I were an objective observer," on a scale ranging from "never do that" (0) to "always do that" (6).
Change in Surface Electromyography RMS and RMS peak time | Change from Baseline to 8-Week Follow-Up
  articipants will undergo sEMG to evaluate the function of the anterior tibialis and lateral gastrocnemius muscles which have been shown to be dysfunctional in patients with L5 and S1 nerve root compression.6,7,72 Measurement will be taken bilaterally, but analyses will be done to compare the symptomatic and asymptomatic side in patients with only unilateral symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Courtney "Katie" Pickworth, ND, MS, Principal Investigator — National University of Natural Medicine
Locations (1):
- National University of Natural Medicine Helfgott Research Institute, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided